CLINICAL TRIAL: NCT04759079
Title: The Effects of Acupuncture Against Postoperative Nausea and Vomit After Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: The Effects of Acupuncture Against Postoperative Nausea and Vomit After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of West Attica (Other)
Responsible Party: Principal Investigator, Theofilos Tsoleridis MD, MA, MSc, PgDip(c), PhD(c), Principal Investigator, University of West Attica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22917
Record Dates: First submitted 2021-02-05; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Postoperative Nausea; Postoperative Vomiting; Laparoscopic Cholecystectomy; Acupuncture
Keywords: Acupuncture; Postoperative Nausea; Postoperative Vomiting; Laparoscopic Cholecystectomy
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Antiemetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture Needles and Antiemetic Drug (Experimental)
  Interventions: Device: Acupuncture Needles; Drug: Antiemetic Drug
- Antiemetic Drug (Active Comparator)
  Interventions: Drug: Antiemetic Drug

INTERVENTIONS:
Device: Acupuncture Needles — Acupuncture Needles placement at the PC6 in association to anti-emetic medication
  Arms: Acupuncture Needles and Antiemetic Drug
Drug: Antiemetic Drug — Administration of Anti-emetic medication without acupuncture

SUMMARY:
Postoperative nausea and vomiting (PONV), represents a common condition after surgery and anesthesia. Acupuncture has been used for centuries for analgesia and quality of life improvement in addition to low cost. This study is a random control trial concerning the antiemetic efficacy of acupuncture associated with intravenous antiemetics in laparoscopic cholecystectomy, in comparison to patients under only antiemetic administration.

One hundred patients were enrolled, regardless of their sex, age, and comorbidity and were randomly allocated in one of two groups. Both anesthesia and antiemetic medication were personalized according to each patient's medical history. In the study group, after anesthesia induction and before pneumoperitoneum application, a sterile stainless steel 0,25 x 25mm acupuncture needle was inserted bilaterally at the PC6 for 20 minutes, rotated manually clockwise and then anticlockwise every 5 minutes and then removed. Fisher's exact test was chosen for statistic evaluation.

There were 8 PONV cases in the study group against 18 cases in the control group. Fisher's exact test highlighted a p-value of P=0,03, marking the difference between the two groups as statistically significant.

Concluding, acupuncture presents a remarkable action against PONV after Laparoscopic Cholecystectomy (LPC). Another remarkable trait of acupuncture is the safety that it offers during application without provoking severe adverse effects. Furthermore, reduced medical costs thanks to decreased postoperative use of antiemetic medication, decreased patients' hospitalization, and reduced re-hospitalization possibility have to be noted. Finally, it has to be mentioned that despite LPC is in general terms painless, the analgesic effects of acupuncture should not be disregarded

ELIGIBILITY:
Inclusion Criteria:

* Adult Male patients undergoing laparoscopic cholecystectomy regardless of other comorbidities.
* Adult Female patients undergoing laparoscopic cholecystectomy regardless of other comorbidities.
* To be able to communicate with personnel.

Exclusion Criteria:

* Patients under 18 years old.
* Inflammation of acupuncture site (PC6).
* Inaccessible acupuncture site (eg. arm amputees, trauma).
* Patients unable to communicate with personnel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
The number of patients of the "acupuncture needles and antiemetic drug" group with postoperative nausea and vomit (PONV), versus the number of patients of the "antiemetic drug" group with PONV. | Immediately after surgery
The number of patients of the "acupuncture needles and antiemetic drug" group with postoperative nausea and vomit (PONV), versus the number of patients of the "antiemetic drug" group with PONV. | 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Rhodes, Rhodes, Dodekanese, Greece

IPD SHARING:
Plan to Share IPD: No